CLINICAL TRIAL: NCT02622685
Title: A Dose Block-randomized, Double-blind, Placebo Controlled, Multiple Dosing, Dose-escalation Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetics of DWP10292 and Ursodeoxycholic Acid in Healthy Male Subjects
Brief Title: A Multiple Dose Study of DWP10292 and UDCA in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: DW_P10292002P
Record Dates: First submitted 2015-04-30; First posted 2015-12-04 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
MeSH Terms: interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- DWP10292 (Experimental): Drug: DWP10292 DWP10292 tablets, oral administration, multiple administration
  Arms: DWP10292
  Interventions: Drug: DWP10292
- DWP10292 Placebo (Placebo Comparator): Drug: Placebo Placebo tablets, oral administration, multiple administrations
  Arms: Placebo
  Interventions: Drug: DWP10292 Placebo
- Ursodeoxycholic acid (UDCA) (Experimental): Drug: Ursodeoxycholic acid (UDCA) UDCA tablets, oral administration, multiple administrations
  Arms: Ursodeoxycholic acid (UDCA)
  Interventions: Drug: Ursodeoxycholic acid (UDCA)
- Ursodeoxycholic acid (UDCA) Placebo (Placebo Comparator): Drug: Placebo Placebo tablets, oral administration, multiple administrations
  Arms: Placebo
  Interventions: Drug: UDCA Placebo

INTERVENTIONS:
Drug: DWP10292 — Drug: DWP10292 tablets, oral administration, multiple administration
  Arms: DWP10292
Drug: DWP10292 Placebo — Placebo tablets, oral administration, multiple administrations
  Arms: DWP10292 Placebo
Drug: Ursodeoxycholic acid (UDCA) — Drug: Ursodeoxycholic acid (UDCA) tablets, oral administration, multiple administration
  Arms: Ursodeoxycholic acid (UDCA)
Drug: UDCA Placebo — Placebo tablets, oral administration, multiple administrations
  Arms: Ursodeoxycholic acid (UDCA) Placebo

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, pharmacokinetics and pharmacodynamics of DWP10292 and UDCA in healthy male volunteers after multiple-dosing.

DETAILED DESCRIPTION:
This study is dose block-randomized, double-blind, placebo controlled, multiple-dosing, dose escalation clinical trial to investigate the safety, tolerability and pharmacokinetic characteristics of DWP 10292 after oral administration in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* A subject who provided written informed consent to participate in this study and cooperative with regard to compliance with study related constraints
* Healthy adult male subjects aged 19 to 45 years
* The subject has a Body weight ≥ 60 kg and < 90 kg and Body Mass Index(BMI) ≥ 18.5 kg/m2 and < 27.0 kg/m2
* A Subject who was judged to be healthy by the investigator to participate in this study based on screening results (according to standard reference index updated recently)

Exclusion Criteria:

* A subject with sign or symptoms or previously diagnosed disease of liver (viral hepatitis), digestive system, cardiovascular, kidney, respiratory, endocrinology, neurology, immune system, hematology, and psychology function or other significant diseases and history or suspicion of current drug abuse and alcohol abuse
* A subject who shows vital signs with the number of systolic blood pressure of ≥140 mmHg or ≤100 mmHg, and the number of diastolic blood pressure of ≥90mmHg or ≤60mmHg
* A subject who donates his blood (whole blood donation within last 2 months or plasma donation within last 1 month) or received a blood transfusion within last 1 month
* Subject who has taken other clinical or licensed medication from another clinical trial within an 3-month period prior to the first administration of the study medication (The last administration of the medication is considered as an end point of the previous clinical trial)
* Subject who smokes an average of 10 cigarettes/day and is unable to quit smoking during the clinical trial

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetics | Multiple blood sample will be collected for 24 hours after last dosing in each of the periods
  Peak Plasma Concentration (Cmax)
Composite of Pharmacokinetics | Multiple blood sample will be collected for 24 hours after last dosing in each of the periods
  Area under the plasma concentration versus time curve (AUC)
Composite of Pharmacokinetics | Multiple blood sample will be collected for 24 hours after last dosing in each of the periods
  Mean residence time (MRT)
Composite of Pharmacokinetics | Multiple blood sample will be collected for 24 hours after last dosing in each of the periods
  Accumulation index

SECONDARY OUTCOMES:
[Safety & tolerability] Incidence of adverse events related with drug | 4 weeks
  Adverse events, Physical exam, Vital sign, laboratory (CBC, chemistry, U/A etc)